CLINICAL TRIAL: NCT00782145
Title: HSCT-CHESS to Enhance Hematopoietic Transplant Recovery
Brief Title: A Web-Based Stem Cell Transplant Support System or Standard Care in Young Patients Undergoing Stem Cell Transplant and Their Families
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Susan Kenyon Parsons, Tufts Medical Center Cancer Center
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: CDR0000613668; R01CA119196 (NIH); TUFTS-8338; WCCC--2007-1357; CHW-07237; CHW-GC-580; DFCI-08-106; CHNMC-08009; CCHMC-0002988; FHCRC-2210
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neuroblastoma; Ovarian Cancer; Psychosocial Effects of Cancer and Its Treatment; Sarcoma
Keywords: psychosocial effects of cancer and its treatment; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; accelerated phase chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; juvenile myelomonocytic leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; childhood myelodysplastic syndromes; primary myelofibrosis; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated childhood rhabdomyosarcoma; previously treated myelodysplastic syndromes; recurrent childhood rhabdomyosarcoma; recurrent neuroblastoma; recurrent ovarian germ cell tumor; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Recurrence; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Primary Myelofibrosis | interventions — Early Intervention, Educational; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Each dyad receives institution-specific care for 6 months, which typically includes psychosocial support for the HSCT recipient and individualized or group education and support for the accompanying parent during the peri-transplant period. They also receive the Web-based Hematopoietic Stem Cell Transplantation (HSCT-) Comprehensive Health Enhancement Support System (HSCT-CHESS) intervention for 6 months. Accompanying parents also identify a companion to receive access to the HSCT-CHESS Web Site.
  The HSCT-CHESS Web site provides ready access to accurate information and resources about pediatric HSCT, practical tips, organizational tools, and other supporting services for use during the transplant process. In addition to collecting data for later analysis, the Web site tracking system allows for further tailoring of information and support for the user, principally by time post transplant.
  Interventions: Other: educational intervention; Other: informational intervention; Other: internet-based intervention; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Other: survey administration; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment; Procedure: standard follow-up care
- Arm II (Active Comparator): Each dyad receives institution-specific usual care for 6 months as described in arm I. Accompanying parents also receive a book from the Blood and Marrow Transplant Information Network (BMT Infonet).
  Interventions: Other: educational intervention; Other: informational intervention; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Other: survey administration; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment; Procedure: standard follow-up care

INTERVENTIONS:
Other: educational intervention
Other: informational intervention
Other: internet-based intervention
  Arms: Arm I
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Other: survey administration
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment
Procedure: standard follow-up care

SUMMARY:
RATIONALE: A Web site for stem cell transplant health information and support may be effective in helping parents improve their health-related knowledge, skills, and quality of life, which may also improve their children's quality of life.

PURPOSE: This randomized phase III trial is studying a Web-based stem cell transplant support system to see how well it works compared with standard care in families of young patients undergoing a stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the ability of a Web-based Hematopoietic Stem Cell Transplantation (HSCT-) Comprehensive Health Enhancement Support System (HSCT-CHESS) to mitigate the impact of a child's HSCT on the health-related quality of life, family functioning, knowledge, skills, and processes of care of the accompanying parent.

Secondary

* To explore the potential mechanisms of action of HSCT-CHESS in improving outcomes in these parents, in terms of parental activation, social support and/or coping skills.
* To explore the impact of HSCT-CHESS on the health-related quality of life of the pediatric HSCT patient, as reported by the parent and child.

OUTLINE: This is a multicenter study. Pediatric hematopoietic stem cell transplantation (HSCT) recipients (ages 2 months-18 years) and accompanying parents are asked to complete a baseline assessment battery by the start of transplant conditioning (the 'run-in' period). If either member of the participating dyad fails to complete all study measures* during this time period, the dyad is withdrawn from the study. The dyads are randomized into 1 of 2 intervention arms.

NOTE: *Measures will not be collected from pediatric patients under 5 years of age at baseline or follow-up.

* Arm I: Each dyad receives institution-specific usual care for 6 months, which typically includes psychosocial support for the HSCT recipient and individualized or group education and support for the accompanying parent during the peri-transplant period. They also receive the Web-based Hematopoietic Stem Cell Transplantation (HSCT-) Comprehensive Health Enhancement Support System (HSCT-CHESS) intervention for 6 months. Accompanying parents also may identify a companion to receive access to the HSCT-CHESS Web site.

The HSCT-CHESS Web site provides ready access to accurate information and resources about pediatric HSCT, practical tips, organizational tools, and other supportive services for use during the transplant process. While the Web site is designed primarily for use by the accompanying parent, it also includes some resources for child and adolescent HSCT recipients that the parent may choose to share. In addition to collecting data for later analysis, the Web site tracking system allows for further tailoring of information and support for the user, principally by time post transplant.

* Arm II: Each dyad receives institution-specific usual care for 6 months as described in arm I. Accompanying parents also receive a book from the Blood and Marrow Transplant Information Network (BMT InfoNet).

Each dyad completes quality-of-life assessment (Child Health Ratings Inventory [CHRIs]-General and CHRIs-HSCT) at day 45, and at 3, 6, 9, and 12 months and CHRIS-General at baseline. The accompanying parent provides demographic information at baseline and 6 months and completes Patient Health Questionnaire (PHQ-9) for depression screening at baseline and 6 and 9 months. The accompanying parent also completes other measures for family and individual coping, social support, process of care, and Internet use at baseline and 6 and 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Disease indications for hematopoietic stem cell transplantation (HSCT)

  * All transplant types allowed
* Scheduled to receive HSCT within the next 30 days

PATIENT CHARACTERISTICS:

* Dyad consisting of age-eligible child and parent
* Child patient with an "accompanying parent" who consents to participate

  * "Accompanying parent" is defined as the parent/legal guardian who physically stays with the recipient during the initial HSCT hospitalization and plans to be present during the follow-up assessments

    * If the responsibility for care giving is shared, parents will designate who will participate (i.e., as study participant)

      * No substitutions are permitted once this decision has been made
  * Accompanying parent must be ≥ 18 years old
* Possesses a working knowledge of English
* Able to sign consent/assent to participate

PRIOR CONCURRENT THERAPY:

* No concurrent participation in another quality-of-life intervention study

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Effect of the Hematopoietic Stem Cell Transplantation Comprehensive Health Enhancement Support System (HSCT-CHESS) on health-related quality of life of the accompanying parent at study entry, day 45 and 3, 6, 9, and 12 months
Effect of HSCT-CHESS on family functioning as reported by the accompanying parent at study entry, 6, and 9 months
Effect of HSCT-CHESS on accompanying parent's knowledge and skills in caring for self and the HSCT recipient, increased confidence interacting with health care provider(s) and greater healthcare participation at study entry, 6, and 9 months

SECONDARY OUTCOMES:
Potential mechanisms of action of HSCT-CHESS in improving parental activation, social support and/or coping skills at study entry and 6 and 9 months
Health-related quality of life of the patient as reported by both parent and child at study entry, day 45, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan K. Parsons, MD, MRP, Principal Investigator — Tufts Medical Center Cancer Center
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin